CLINICAL TRIAL: NCT02581501
Title: Prospective Phase I Study of Gax (Gemcitabine, ABRAXANE, and Xeloda) for Metastatic Pancreatic Cancer Protocol # TSH - APG - 2015-01
Brief Title: Prospective Phase I Study of GAX for Metastatic Pancreatic Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to no enrollment, Celgene (sponsor) withdrew funding
Sponsor: Stamford Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: StamfordH
Record Dates: First submitted 2015-10-19; First posted 2015-10-21 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Pancreatic Cancer
Keywords: Xeloda; Gemcitabine; Abraxane; Pancreatic Cancer; Metastatic Cancer; Phase I; 5-FU; Capecitabine; Gemzar; NAB-Paclitaxel; Chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — Albumin-Bound Paclitaxel; Capecitabine; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine, ABRAXANE®, and Xeloda (Experimental): Level-1
  ABRAXANE® 75 mg/m2 over 30 min Days 5 and 12
  GEMCITABINE 600 mg/m2 over 60 min Days 5 and 12.
  XELODA 500 mg/m2 BID D 1-14 capped at total dose of 2000 mg/day
  Level 1
  ABRAXANE® 100 mg/m2 over 30 min Days 5 and 12
  GEMCITABINE 600 mg/m2 over 60 min Days 5 and 12
  XELODA 500 mg/m2 BID D 1-14 capped at total dose of 2000 mg/day
  Level 2
  ABRAXANE® 125 mg/m2 over 30 min Days 5 and 12
  GEMCITABINE 600 mg/m2 over 75 min Days 5 and 12
  XELODA 500 mg/m2 BID D 1-14 capped at total dose of 2000 mg/day
  Level 3
  ABRAXANE® 125 mg/m2 over 30 min Days 5 and 12
  GEMCITABINE 750 mg/m2 over 75 min Days 5 and 12
  XELODA 500 mg/m2 BID D 1-14 capped at total dose of 2000 mg/day
  Interventions: Drug: GAX - Gemcitabine, Abraxane and Xeloda

INTERVENTIONS:
Drug: GAX - Gemcitabine, Abraxane and Xeloda — GAX represents a novel approach to the development of cancer chemotherapy agents in pancreatic cancer and is based upon extensive laboratory investigations for the induction of apoptosis in pancreatic carcinoma cells. It is our expectation that this combination will induce apoptotic pathways downstream of biochemical mechanisms of resistance and synergistically induce pathways for apoptosis that are non-p53 dependent, which have not been previously explored in chemotherapy trials for this cancer.
  Other Names: Chemotherapy, Pancreatic Cancer

SUMMARY:
GAX represents a novel approach to the development of cancer chemotherapy agents in pancreatic cancer and is based upon extensive laboratory investigations for the induction of apoptosis in pancreatic carcinoma cells.

DETAILED DESCRIPTION:
It is the investigators expectation that this combination will induce apoptotic pathways downstream of biochemical mechanisms of resistance and synergistically induce pathways for apoptosis that are non-p53 dependent, which have not been previously explored in chemotherapy trials for this cancer. ABRAXANE® is novel in that it induces apoptosis to the same degree in mutant and wt p53 cancers. Mutant p53 tumors occur in 80-90% of PC and mutant p53 is thought of as one of the major mechanisms of drug resistance.

Furthermore, the investigators will be starting Xeloda and gemcitabine at slightly lower doses than the initial GTX studies. This is because the investigators have found that the efficacy is maintained at these slightly lower doses while side effects are minimized. The reason that GTX works at lower doses, as well as higher doses, is the synergy between drugs. Drug regimens that are synergistic can maintain their antitumor effect at doses lower than in non-synergistic regimens, but must maintain their dose intensity to achieve their anti-tumor effect. RECIST 1.1 criteria will be utilized for judging response, progression and stable disease. Overall assessment of the data will be by intention to treat analysis (ITT).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of pancreas metastatic to any distant site. (Stage IV).
2. Must have a lesion reproducibly measurable by CT or MRI scans per Recist 1.1 criteria
3. Prior radiation and surgery allowed (except Target lesions) but GAX treatment should be: >3 weeks since major surgery

   1. Bilirubin < 1.5 mg/dL
   2. Patients must have adequate liver function: AST and ALT < 2.5 X upper limit of normal, alkaline phosphatase < 2.5 X upper limit of normal, unless bone metastasis is present (<5 X upper limit of normal) in the absence of liver metastasis.
   3. Patients must have adequate bone marrow function: Platelets >100,000, Hemoglobin > 9.0g/dL and ANC > 1,500
   4. Patients must have adequate renal function: creatinine <1.5 mg/dL is recommended
4. Women of childbearing potential and sexually active males must use an effective contraception method during treatment and for three months after completing treatment.
5. Patients must have < Grade 2 pre-existing peripheral neuropathy (per CTCAE)
6. Clinical Parameters Life expectancy > three months Age ≥ 18 years and ≤ 75 years Performance status 0-1 (ECOG) Pre-existing Peripheral Neuropathy (sensory) must be ˂ grade 2 Able to tolerate oral medications
7. Informed Consent: Each patient must be completely aware of the nature of his/her disease process and must willingly give consent after being informed of the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks, and discomforts.
8. PT/PTT within normal or therapeutic limits as determined by the investigator. All subjects will be on Xeloda, use of warfarin is exclusionary.

Exclusion Criteria:

1. Neuroendocrine cancer should be ruled out by histology or immunohistochemical staining of the specimen. Mixed histology, pancreatic neuroendocrine and adenocarcinoma tumors, will also be excluded.
2. Prior chemotherapy is allowed, as long as less than or equal to two of the components of GAX were used previously for their treatment: this includes gemcitabine, capecitabine, 5-FU, or ABRAXANE® .
3. Hypersensitivity: Patients with a history of severe hypersensitivity reaction to taxanes or other drugs formulated with polysorbate 80, or any of the other drugs in the GAX regimen are excluded.
4. Serious medical or psychiatric illness preventing informed consent or intensive treatment (e.g. serious infection) that would in the opinion of the investigator, increase the risk of serious neutropenic complications.
5. Serious medical risk factors involving any of the major organ systems, or serious psychiatric disorders, which could compromise the subject's safety or the study data integrity.
6. Patients with compromised immune systems who are at increased risk of toxicity and lethal infections when treated with marrow-suppressive therapy.
7. Serious cardiovascular thromboembolic disease, including: congestive heart failure NYHA class III or greater; unstable angina or new onset angina (starting within three months of screening for this protocol), or myocardial infarction within the past 3 months (prior to screening); serious cardiac arrhythmias requiring therapy; cerebrovascular accident including transient ischemic attacks within the past 3 months (prior to screening).
8. Serious non-healing wound, ulcer, or bone fracture.
9. Evidence or history of bleeding diathesis.
10. Major surgery, open biopsy or significant traumatic injury within 3 weeks of receiving first study drug.
11. Use of cytochrome P450 enzyme inducing drugs such as: antiepileptic drugs (phenytoin, carbamazepine, or phenobarbital, but not Keppra), or St. John's Wort or rifampin (rifampicin).
12. Prior malignancy in last 2 years other than curatively treated carcinoma in-situ of any site, non-melanoma skin cancer, or Stage I breast and/or bladder cancers (in situ), or early stage prostate cancer Stage I or II, curatively treated by surgery and/or radiation.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Identification of Maximum Tolerated Dose and Dose Intensity in Patients with Pancreatic Cancer | 24 months
  To determine the dose for Phase II study - identification of the maximum tolerated dose (MTD) and dose intensity in patients with advanced pancreatic cancer. As a Phase I study, primary objective is toxicity identification, not treatment efficacy.

SECONDARY OUTCOMES:
Progression Free Survival | 6 years
  To evaluate the response rate (using RECIST 1.1 criteria), the Progression free survival (PFS) and Overall Survival (OS) with treatment.

OTHER OUTCOMES:
Assess Safety and Toxicity based upon NCI Common toxicity criteria version 4.1. | 24 Months
  To assess the safety and toxicities to this regimen based upon NCI Common toxicity criteria version 4.1.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Gulati, M.D, Principal Investigator — Stamford Hospital
Locations (1):
- Stamford Hospital Bennett Cancer Center, Stamford, Connecticut, United States